CLINICAL TRIAL: NCT02855190
Title: Pilot Comparative Study of PET/MR and PET/CT With Different Tracers (18F-FDG and 68Gallium Citrate) in the Diagnosis of Periprosthetic Joint Infection
Brief Title: Comparative Study With Different Tracers (18F-FDG and 68Gallium Citrate) in the Diagnosis of Periprosthetic Joint Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzu-Chen Yen, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 103-7226A
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Infection and Inflammatory Reaction Due to Internal Joint Prosthesis
Keywords: Ga68-citrate; FDG; PET/MR and PET/CT; Periprosthetic joint infection
MeSH Terms: conditions — Infections | interventions — gallium citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-citrate and 18F-FDG PET scans (Experimental): The recruited subject with surgery/pathology proved periprosthetic joint infection will undergo total four PET scans at two different stages. At first stage, subsequent FDG PET/CT and Ga68 citrate PET/CT scans on different two days will be arranged before infective prosthesis is removed. Eight to twelve weeks after the 1st stage operation, patient will receive two subsequent PET/MR scans using Ga-68 Citrate and FDG on different two days, respectively. For the subject without surgery/pathology proved infection, PET/MR scans will NOT be applied.
  Interventions: Other: 68Ga-citrate and 18F-FDG PET scans

INTERVENTIONS:
Other: 68Ga-citrate and 18F-FDG PET scans — 68Ga-citrate and 18F-FDG PET/CT or PET/MR scans before operations

SUMMARY:
This is an open-labelled two-arm pilot comparative prospective study. All the subjects will undergo image assessment in the two stages of exchange arthroplasty surgery. At the first stage, each enrolled subject will receive both FDG and Ga68 citrate PET/CT scans before the first operation for periprosthetic Joint Infection (PJI). Thus, the test results of FDG and Ga68 for each individual can be obtained. After the first operation, the surgery/biopsy proof can be obtained as the gold standard. The subjects those with PJI negative will complete the process at the first stage.

And the second stage of this study will be based on the subjects with positive PJI from the first operation. They will receive both FDG and Ga68 citrate PET/MR scans after antibiotic bone cement was implanted. The sensitivity/accuracy of the two tracers for PET/MR can be calculated and compared. This stage is aimed to answer whether PET/MR scan is a feasible imaging tool to provide diagnostic information of infection control status after the resection arthroplasty of hip/knee PJIs, especially with the implantation of antibiotic loaded bone cement.

In the second stage, the investigators shift the imaging modality to PET/MR based on the following reasons: (1) MRI itself has no radiation burden; (2) MRI provides more accurate tissue contrast information and therefore better anatomic delineation; and (3) currently there was no study indicating the existence of ABLC may hamper the interpretation of images.

The study duration is expected to be completed in a period of 3 year. It plans to enrol a total of 40 evaluable subjects with suspicious. And we expect the PJI prevalence will be around 75%, i.e. the anticipated number of subjects of true PJI is around 30. The sample size and the prevanence is given based on the clinical availability and consideration.

DETAILED DESCRIPTION:
The recruited subject subject with periprosthetic joint infection will undergo total four PET scans at two different stages. At first stage, subsequent FDG PET/CT and Ga68 citrate PET/CT scans on different two days will be arranged before infective prosthesis is removed. Eight to twelve weeks after the 1st stage operation, patient will receive two subsequent PET/MR scans using Ga-68 Citrate and FDG on different two days, respectively. The PET images will be visually examined by a nuclear medicine physician and will be reported if any abnormal uptake higher than background by their location and standard uptake value (SUV). The CT/MR images will be reported by a radiologist using standard reading procedures, respectively. The lesions on the PET scan will be correlated to the computed tomography and magnetic resonance images, and the final sensitivity, specificity, and accuracy will be calculated according to the histopathology results or composite clinical and laboratory data.

On the scan day using Ga68-Citrate, baseline electrocardiogram, complete blood count (CBC), and biochemistry profiles including serum alanine transaminase (ALT) and creatinine (Cre) level will be done prior to injection of the radio-pharmaceutical (Ga68-Citrate). Vital signs will be measured before the scan beginning. After completing exam, the electrocardiogram and vital signs will be measure again, and the subject will be released if there is no discomfort. The subject will return to the clinic within 1 week after Ga68-citrate scan. CBC, biochemistry profiles will be checked again for safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically-proved or -suspicious periprosthetic joint infection and treated with two-stage exchange arthroplasty
2. Age equals or more than 20 years old
3. Willing to sign the informed consent

Exclusion Criteria:

1. Unable to tolerate PET/MR or PET/CT scan, such as those with magnetic implants (e.g. those received intracranial aneurysm surgery, cardiac pacemaker, artificial valves replacement, artificial ears), renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), claustrophobia, unable to lie still, allergy to medium contrast.
2. Unable to give informed consent
3. Patient who is pregnant or lactating
4. Unwilling to use contraceptives during nuclide medicine examinations.
5. Allergy history to FDG or Ga68-citrate, significant abnormal lab data, and high risk to conduct examination after evaluations of PI.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of the two PET/CT tracers (18F-FDG and 68Gallium citrate) in detecting periprosthetic joint infection | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yen Tzu-Chen, MD,PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bauman G, Belhocine T, Kovacs M, Ward A, Beheshti M, Rachinsky I. 18F-fluorocholine for prostate cancer imaging: a systematic review of the literature. Prostate Cancer Prostatic Dis. 2012 Mar;15(1):45-55. doi: 10.1038/pcan.2011.35. Epub 2011 Aug 16. PMID 21844889
- [Result] Mohler JL, Armstrong AJ, Bahnson RR, Boston B, Busby JE, D'Amico AV, Eastham JA, Enke CA, Farrington T, Higano CS, Horwitz EM, Kantoff PW, Kawachi MH, Kuettel M, Lee RJ, MacVicar GR, Malcolm AW, Miller D, Plimack ER, Pow-Sang JM, Roach M 3rd, Rohren E, Rosenfeld S, Srinivas S, Strope SA, Tward J, Twardowski P, Walsh PC, Ho M, Shead DA. Prostate cancer, Version 3.2012: featured updates to the NCCN guidelines. J Natl Compr Canc Netw. 2012 Sep;10(9):1081-7. doi: 10.6004/jnccn.2012.0114. PMID 22956807
- [Result] Picchio M, Castellucci P. Clinical Indications of C-Choline PET/CT in Prostate Cancer Patients with Biochemical Relapse. Theranostics. 2012;2(3):313-7. doi: 10.7150/thno.4007. Epub 2012 Mar 12. PMID 22448197
- [Result] Schwarzenbock S, Souvatzoglou M, Krause BJ. Choline PET and PET/CT in Primary Diagnosis and Staging of Prostate Cancer. Theranostics. 2012;2(3):318-30. doi: 10.7150/thno.4008. Epub 2012 Mar 15. PMID 22448198
- [Result] Beer AJ, Eiber M, Souvatzoglou M, Schwaiger M, Krause BJ. Radionuclide and hybrid imaging of recurrent prostate cancer. Lancet Oncol. 2011 Feb;12(2):181-91. doi: 10.1016/S1470-2045(10)70103-0. Epub 2010 Jul 6. PMID 20599424
- [Result] Umbehr MH, Muntener M, Hany T, Sulser T, Bachmann LM. The role of 11C-choline and 18F-fluorocholine positron emission tomography (PET) and PET/CT in prostate cancer: a systematic review and meta-analysis. Eur Urol. 2013 Jul;64(1):106-17. doi: 10.1016/j.eururo.2013.04.019. Epub 2013 Apr 19. PMID 23628493
- [Result] Wetter A, Lipponer C, Nensa F, Beiderwellen K, Olbricht T, Rubben H, Bockisch A, Schlosser T, Heusner TA, Lauenstein TC. Simultaneous 18F choline positron emission tomography/magnetic resonance imaging of the prostate: initial results. Invest Radiol. 2013 May;48(5):256-62. doi: 10.1097/RLI.0b013e318282c654. PMID 23462678
- [Result] Abuzallouf S, Dayes I, Lukka H. Baseline staging of newly diagnosed prostate cancer: a summary of the literature. J Urol. 2004 Jun;171(6 Pt 1):2122-7. doi: 10.1097/01.ju.0000123981.03084.06. PMID 15126770
- [Result] Souvatzoglou M, Eiber M, Martinez-Moeller A, Furst S, Holzapfel K, Maurer T, Ziegler S, Nekolla S, Schwaiger M, Beer AJ. PET/MR in prostate cancer: technical aspects and potential diagnostic value. Eur J Nucl Med Mol Imaging. 2013 Jul;40 Suppl 1:S79-88. doi: 10.1007/s00259-013-2445-4. Epub 2013 May 24. PMID 23703457
- [Derived] Tseng JR, Chang YH, Yang LY, Wu CT, Chen SY, Wan CH, Hsiao IT, Yen TC. Potential usefulness of 68Ga-citrate PET/CT in detecting infected lower limb prostheses. EJNMMI Res. 2019 Jan 3;9(1):2. doi: 10.1186/s13550-018-0468-3. PMID 30607646